CLINICAL TRIAL: NCT00880672
Title: Apoptosis and Expression of Neovascularization-related Factors in Human Prostate Tissue After Administration of Dutasteride
Brief Title: Effect of Dutasteride on HIF-1alpha and VEGF in the Prostate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: The Korean Urological Association (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Ja Hyeon Ku,, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHKu1
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2009-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: prostate, dutasteride; vascular endothelial growth factor; hypoxia inducible factor
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dutasteride (Active Comparator): oral, 5mg, once per day, 2 weeks
  Interventions: Drug: dutasteride
- placebo (Placebo Comparator): oral, 5mg, once per day, 2 weeks

INTERVENTIONS:
Drug: dutasteride — 5mg, oral, daily, 2-4 weeks
  Arms: dutasteride

SUMMARY:
The purpose of this study is to determine whether dutasteride may influence the expression of angiogenesis factors such as hypoxia inducible factor (HIF)-1alpha and vascular endothelial growth factor (VEGF) in patients with lower urinary tract symptoms/benign prostatic hyperplasia (LUTS/BPH).

DETAILED DESCRIPTION:
A total of 41 patients awaiting transurethral resection of the prostate (TURP) will be divided into two groups (1:1); twenty patients will receive no medication and 21 will receive 0.5 mg dutasteride daily for 2 to 4 weeks until TURP. In both groups, the extent, intensity and intracellular location of hypoxia inducible factor (HIF)-1alpha and vascular endothelial growth factor (VEGF)will be evaluated. Microvessel density will be also compared in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* 50 years old or older
* International Prostate Symptom Score (IPSS) >8
* Maximum flow rate (Qmax) <15 ml/s
* transurethral resection of the prostate (TURP)

Exclusion Criteria:

* urethral catheter
* urinary tract infection (UTI)
* liver disease
* renal disease
* unexplained hematuria
* prostate specific antigen (PSA) > 4ng/ml (included if prostate biopsy was negative)
* interstitial cystitis
* bladder cancer or prostate cancer
* pelvic surgery or irradiation

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
HIF-1a and VEGF expression | 2 weeks
  effects of dutasteride on the expression of angiogenesis markers in rat and human prostates

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Seung paick, MD, PhD, Principal Investigator — Dept. of Urology, Seoul National University Hospital